CLINICAL TRIAL: NCT04527666
Title: Anticoagulation Treatment of Patients With Gastroesophageal Varices and JAK2 V617 Mutation
Brief Title: Anticoagulation in Gastroesophageal Varices and JAK2 Mutation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, XiaoquanHUANG, Resident, Shanghai Zhongshan Hospital
Other Study IDs: ZS-ANTICO-JAK2
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Varices; JAK2 Mutation; Myeloproliferative Neoplasm
Keywords: portal hypertension; gastroesophageal varices; jak2 mutation; myeloproliferative neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders; Hypertension, Portal | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anticoagulation group: Patients with JAK2 mutation and gastroesophageal varices receive anticoagulation agents.
  Interventions: Drug: Anticoagulation Agents
- Control group: Patients with JAK2 mutation and gastroesophageal varices who didn't receive anticoagulation agents.

INTERVENTIONS:
Drug: Anticoagulation Agents — Patients receive anticoagulation agents including low molecular weight heparin, warfarin, rivaroxaban, et al.
  Groups: Anticoagulation group

SUMMARY:
Myeloproliferative neoplasms (MPNs), including polycythemia vera, essential thrombocythemia, and primary myelofibrosis, may lead to gastroesophageal varices. The quality of life, morbidity, and mortality of MPN patients mainly depend on disease-related symptoms, thromboembolic and hemorrhagic complications. Previous studies have shown that JAK2 V617F has a prominent role in vascular risk and MPN-associated gastroesophageal varices. The aim of this study is to evaluate the efficacy of anticoagulation in patients with JAK2 mutation and gastroesophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-75
* diagnosed as portal hypertension by contrast-enhanced computed tomography
* diagnosed as JAK2 positive

Exclusion Criteria:

* not had portal contrast-enhanced computed tomography
* not had JAK2 mutation test
* other factors judged by the investigator that may affect the safety of the subject or the compliance of the trial. Such as serious illnesses (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric and/or esophageal varices and JAK2 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes of portal vein thrombosis | 1 year
  The changes of portal vein thrombosis including progression, disappear or unchanged.

SECONDARY OUTCOMES:
The occurrence of variceal bleeding | 1 year
  The occurrence of variceal bleeding including haematemesis and melena
Overall survival | 1 year
  Overall survival rate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenfield G, McMullin MF. Splanchnic venous thrombosis in JAK2 V617F mutation positive myeloproliferative neoplasms - long term follow-up of a regional case series. Thromb J. 2018 Dec 19;16:33. doi: 10.1186/s12959-018-0187-z. eCollection 2018. PMID 30574023
- [Background] Yan M, Geyer H, Mesa R, Atallah E, Callum J, Bartoszko J, Yee K, Maganti M, Wong F, Gupta V. Clinical features of patients with Philadelphia-negative myeloproliferative neoplasms complicated by portal hypertension. Clin Lymphoma Myeloma Leuk. 2015 Jan;15(1):e1-5. doi: 10.1016/j.clml.2014.04.004. Epub 2014 Jun 11. PMID 25027569
- [Background] Magaz M, Alvarez-Larran A, Colomer D, Lopez-Guerra M, Garcia-Criado MA, Mezzano G, Belmonte E, Olivas P, Soy G, Cervantes F, Darnell A, Ferrusquia-Acosta J, Baiges A, Turon F, Hernandez-Gea V, Garcia-Pagan JC. Next-generation sequencing in the diagnosis of non-cirrhotic splanchnic vein thrombosis. J Hepatol. 2021 Jan;74(1):89-95. doi: 10.1016/j.jhep.2020.06.045. Epub 2020 Jul 15. PMID 32679300
- [Result] Reilly CR, Babushok DV, Martin K, Spivak JL, Streiff M, Bahirwani R, Mondschein J, Stein B, Moliterno A, Hexner EO. Multicenter analysis of the use of transjugular intrahepatic portosystemic shunt for management of MPN-associated portal hypertension. Am J Hematol. 2017 Sep;92(9):909-914. doi: 10.1002/ajh.24798. Epub 2017 Jul 26. PMID 28543980